CLINICAL TRIAL: NCT02417467
Title: Evaluating the Efficacy of E-Cigarette Use for Smoking Cessation (E3) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Mark Eisenberg, Professor of Medicine, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E3; MOP-133727 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2015-04-01; First posted 2015-04-15 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Smoking Cessation
Keywords: Electronic cigarette; E-cigarette; Smoking cessation
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nicotine E-Cigarette and Counseling (Experimental): As with standard nicotine replacement therapies, participants are expected to self-regulate administration of nicotine e-cigarettes according to their withdrawal symptoms. The manufacturer recommends each vaping session to last approximately 10 puffs, with one puff every 30 seconds over a span of approximately 4.5 minutes.
  Smoking cessation/relapse prevention counselling will be provided for a minimum of 30 minutes at baseline, 10 minutes during telephone follow-ups, and 15 minutes at clinic visits (20 minutes at week 4). Counselling will consist of a number of approaches, including reviewing smoking history, development/revision of a quit plan, encouragement of self-monitoring, review of triggers and challenges, and skill development.
  Interventions: Other: Nicotine E-Cigarette; Behavioral: Counseling
- Non-Nicotine E-Cigarette and Counseling (Other): Participants are expected to self-regulate administration of e-cigarettes. The manufacturer recommends each vaping session to last approximately 10 puffs, with one puff every 30 seconds over a span of approximately 4.5 minutes.
  Smoking cessation/relapse prevention counselling will be provided for a minimum of 30 minutes at baseline, 10 minutes during telephone follow-ups, and 15 minutes at clinic visits (20 minutes at week 4). Counselling will consist of a number of approaches, including reviewing smoking history, development/revision of a quit plan, encouragement of self-monitoring, review of triggers and challenges, and skill development.
  Interventions: Other: Non-Nicotine E-Cigarette; Behavioral: Counseling
- Counseling (Other): Smoking cessation/relapse prevention counselling will be provided for a minimum of 30 minutes at baseline, 10 minutes during telephone follow-ups, and 15 minutes at clinic visits (20 minutes at week 4). Counselling will consist of a number of approaches, including reviewing smoking history, development/revision of a quit plan, encouragement of self-monitoring, review of triggers and challenges, and skill development.
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Other: Nicotine E-Cigarette
  Arms: Nicotine E-Cigarette and Counseling
Other: Non-Nicotine E-Cigarette
  Arms: Non-Nicotine E-Cigarette and Counseling
Behavioral: Counseling

SUMMARY:
Smoking-related diseases contribute to the death of more than 37,000 Canadians annually. Of that number, almost one-third die of cardiovascular-related causes. Smoking cessation can decrease the additional risk of heart disease by 50% after 1 year. However, even using smoking cessation therapies, only 10-20% of smokers will be able to successfully quit smoking long-term. Therefore, new and alternative treatments are needed.

The e-cigarette is a battery-powered device approximately the size and shape of a cigarette that creates a smoke-free vapour which is inhaled by the user. Since it feels like smoking a cigarette, using the e-cigarette may help some smokers quit. Some e-cigarettes also contain nicotine, which can reduce withdrawal symptoms from quitting smoking. However, e-cigarettes have not been approved for use for smoking cessation by Health Canada or the FDA. Despite this, these devices are rising in popularity. A recent US Centers for Disease Control survey found that of smokers who were motivated to quit within the next 6 months, 48.5% had tried e-cigarettes.

The Evaluating the Efficacy of E-Cigarette Use for Smoking Cessation (E3) Trial will be the first large trial to address the important issue of e-cigarettes for smoking cessation in Canada. The trial will randomly assign participants to receive nicotine e-cigarettes and minimal counseling, non-nicotine e-cigarettes and minimal counseling, or only minimal counseling for 12 weeks. Participants will then be followed for one year to see which (if any) group is more likely to have quit or reduced their smoking. Information about potential side effects and safety will also be collected. The E3 Trial will provide law-makers and the public with important information about the use of e-cigarettes for smoking cessation.

DETAILED DESCRIPTION:
I. OVERALL STUDY OBJECTIVE The Evaluating the Efficacy of E-Cigarette use for Smoking Cessation (E3) Trial is a 5-year, multi-centre, randomized controlled trial (RCT) that seeks to assess the efficacy, safety, and tolerability of nicotine and non-nicotine electronic cigarettes (e-cigarettes) for smoking cessation in the general population.

II. SPECIFIC OBJECTIVES

1. To compare the efficacy of nicotine and non-nicotine e-cigarettes used with individual counselling for smoking cessation, to that of individual counselling alone, in terms of biochemically-validated 7-day point prevalence smoking abstinence at 52 weeks.
2. To examine the effect of nicotine and non-nicotine e-cigarettes on other measures of smoking reduction and cessation, including continuous abstinence and daily cigarette consumption at 4, 12, 24, and 52 weeks.
3. To describe the safety and tolerability of nicotine and non-nicotine e-cigarettes in terms of serious adverse events (SAEs), adverse events (AEs), drop-out rates due to side effects, and therapy adherence over the 12 week treatment period.

I. RATIONALE Smoking-related diseases contribute to the death of more than 37,000 Canadians annually. Of that number, almost one-third die of cardiovascular-related causes. Smoking cessation can decrease the additional risk of heart disease by 50% after one year of abstinence. However, even using traditional smoking cessation therapies, only 10-20% of smokers will be able to successfully quit smoking long-term. Therefore, new and alternative treatments are needed. The e-cigarette is a battery-powered device approximately the size and shape of a cigarette that creates a smoke-free vapour that is inhaled by the user, and is available in nicotine and non-nicotine varieties. Its mimicry of the act of smoking gives it the potential to target the habit-forming mechanism of smoking, and to mitigate withdrawal symptoms with nicotine replacement (in the case of nicotine e-cigarettes). However, e-cigarettes have not been approved for use for smoking cessation by Health Canada or the US Food and Drug Administration. Despite this, these devices are rising in popularity. A recent survey found that of smokers motivated to within 6 months, 48.5% had tried e-cigarettes. The E3 Trial will be the first conducted in the general population of Canadian smokers motivated to quit. It will also provide the longest-term (52 weeks) follow-up data on smoking reduction and cessation in smokers motivated to quit with the e-cigarette.

II. METHODS The investigators will conduct a multi-centre RCT with a treatment period of 12 weeks and follow-up of 52 weeks. A total of 486 participants will be randomized to one of three treatment arms: (1) nicotine e-cigarettes with individual counselling, (2) non-nicotine e-cigarettes with individual counselling, or (3) individual counselling alone. Eligible participants will be recruited from the general population, be at least 18 years of age, will self-identify as regular smokers (≥10 cigarettes per day for at least one year), and be motivated to quit. Participants will complete telephone follow-ups at weeks 1, 2, and 8. The participants will also return for clinic visits at weeks 4, 12, 24, and 52. Biochemically-validated smoking abstinence will be measured at all clinic visits using exhaled carbon monoxide. At follow-up calls and visits, the investigators will collect information about self-reported smoking, e-cigarette use, withdrawal symptoms, and side effects. The primary analysis will compare point-prevalence abstinence at 52 weeks between participants randomized to nicotine e-cigarettes versus individual counselling alone. Similar analyses will be conducted to compare abstinence across other trial arms. In secondary analyses, the investigators will examine point-prevalence abstinence at other follow-ups, as well as the effect of treatment group on continuous abstinence, daily cigarette consumption, and the occurrence of clinical events and side effects. A sample size of 486 was identified through power calculation, based on a 52-week point prevalence abstinence rate of 10% among participants randomized to counselling, with >80% power to detect a ≥12% absolute difference in the prevalence of smoking abstinence at 52 weeks (e.g., a prevalence of abstinence in the nicotine e-cigarette group of 22%) with a two-tailed α of 0.05.

III. SIGNIFICANCE E-cigarettes are popular devices that may have the potential to facilitate smoking cessation. The E3 Trial will provide regulators, health care professionals, and smokers with important information about the efficacy and safety of e-cigarettes for smoking cessation.

IV. ADDENDUM The primary endpoint was changed from 52 weeks to 12 weeks following the early termination of enrollment (77% of target enrollment) due to a delay in product manufacturing.

ELIGIBILITY:
Inclusion Criteria:

* Active smoker, 10 or more cigarettes per day, on average, for the past year;
* Age of 18 years or older;
* Motivated to quit according to the Motivation To Stop Scale (MTSS) (level 5 or higher);
* Able to understand and to provide informed consent in English or French;
* Likely to be available for follow-up (1 year).

Exclusion Criteria:

* Medical condition with a prognosis < 1 year;
* Current or recent cancer (less than 1 year in remission);
* Pregnant or lactating females;
* Current or recent use (in the past 30 days) of any pharmacotherapy or behavioural therapy for smoking cessation (e.g., Nicotine Replacement Therapies, bupropion, varenicline, or counseling);
* Any e-cigarette use (nicotine or non-nicotine) in the past 60 days, or ever use of any e-cigarette for more than 7 days consecutively;
* History of psychosis, schizophrenia, or bipolar disorder;
* Less than one month following a myocardial infarction, life-threatening arrhythmia, severe or worsening angina pectoris, or cerebral vascular accident;
* Use of any illegal drugs in the past year (excluding marijuana);
* Planned use of tobacco products other than conventional cigarettes (e.g., cigarillos, cigars, snuff, shisha, etc.) or marijuana during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2016-11; Primary Completion 2019-12 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with 7-day point prevalence smoking abstinence | 52 weeks
  The primary outcome measure is 7-day point prevalence smoking abstinence at 52 weeks. Smoking abstinence for this measure is defined as self-report smoking abstinence for the previous 7 days, and a measurement of exhaled carbon monoxide less than 11 ppm, at 52 weeks.
  The primary end point will be analyzed on an intention-to-treat (ITT) basis.This ITT analysis assumes that those who withdrew consent or were lost to follow-up had returned to smoking at their baseline rates. This assumption is common in smoking cessation trials.

SECONDARY OUTCOMES:
Number of participants with 7-day point prevalence smoking abstinence | 4, 12, and 24 weeks
  Biochemically-validated 7-day point prevalence smoking abstinence at 4, 12 and 24 weeks, defined as self-reported abstinence in the past 7 days with exhaled carbon monoxide less than 11 ppm.
Number of participants with continuous abstinence from smoking | 4, 12, 24, and 52 weeks
  Biochemically-validated continuous abstinence at 4, 12, 24, and 52 weeks, defined as self-reported abstinence since baseline with exhaled carbon monoxide less than 11 ppm at all follow-up clinic visits.
Change in daily cigarette consumption | 1, 2, 4, 8, 12, 18, 24, and 52 weeks
  Change in self-reported mean number of daily conventional cigarette consumption from baseline to weeks 1, 2, 4, 8, 12, 18, 24, and 52.
The frequency of serious adverse events | 12 weeks
  The number of serious adverse events (SAE) reported over the 12 week treatment period.
  A SAE is defined as an adverse event which requires in-patient hospitalization or prolongation of existing hospitalization, that causes congenital malformation, that results in persistent or significant disability or incapacity, that is life-threatening, or that results in death.
  These SAEs will be reported to the Institutional Review Board, a Data and Safety Monitoring Board (DSMB), and Health Canada, as appropriate. The DSMB will provide oversight of safety and will establish stopping criteria for the trial at their first meeting. An Endpoints Evaluation Committee will be responsible for the evaluation and classification of all SAEs.
The frequency of adverse events | 12 weeks
  The number of adverse events reported over the 12 week treatment period. An adverse event is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the trial drug, whether or not considered related to the e-cigarettes.
The frequency of drop-outs | 12 weeks
  The number of drop-outs due to side effects of the e-cigarettes over the 12 week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Eisenberg, MD MPH, Principal Investigator — McGill University, Jewish General Hospital
Locations (16):
- Canada (16):
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Allen Greenspoon Medicine Profesionnal Corporation, Hamilton, Ontario
  - Baran Medicine Professional Corporation, Kingston, Ontario
  - Institut de recherche de l'Hôpital Montfort, Ottawa, Ontario
  - The Bridge Engagement Centre, Ottawa, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Canadian Centre for Clinical Trials, Thornhill, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Hôpital Cité-de-la-Santé, Laval, Quebec
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Institut de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Quebec
  - Centre de recherche sur le vieillissement, Sherbrooke, Quebec

REFERENCES:
- [Derived] Lyzwinski L, Dong M, Wolfinger RD, Filion KB, Eisenberg MJ. e-Cigarettes, Smoking Cessation, and Weight Change: Retrospective Secondary Analysis of the Evaluating the Efficacy of e-Cigarette Use for Smoking Cessation Trial. JMIR Public Health Surveill. 2024 Sep 16;10:e58260. doi: 10.2196/58260. PMID 39283667
- [Derived] Prell C, Hebert-Losier A, Filion KB, Reynier P, Eisenberg MJ. Evaluating the impact of varying expired carbon monoxide thresholds on smoking relapse identification: insights from the E3 trial on e-cigarette efficacy for smoking cessation. BMJ Open. 2023 Oct 13;13(10):e071099. doi: 10.1136/bmjopen-2022-071099. PMID 37832989
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Eisenberg MJ, Hebert-Losier A, Windle SB, Greenspoon T, Brandys T, Fulop T, Nguyen T, Elkouri S, Montigny M, Wilderman I, Bertrand OF, Bostwick JA, Abrahamson J, Lacasse Y, Pakhale S, Cabaussel J, Filion KB; E3 Investigators. Effect of e-Cigarettes Plus Counseling vs Counseling Alone on Smoking Cessation: A Randomized Clinical Trial. JAMA. 2020 Nov 10;324(18):1844-1854. doi: 10.1001/jama.2020.18889. PMID 33170240